CLINICAL TRIAL: NCT02533752
Title: Canadian WATCHMAN Registry
Acronym: WATCHMAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiology Research UBC (Other)
Responsible Party: Principal Investigator, Jacqueline Saw, MD, Research Director, Cardiology Research UBC
Other Study IDs: H14-01816
Record Dates: First submitted 2015-03-24; First posted 2015-08-27 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
Keywords: Left Atrial Appendage Closure; Watchman device; LAA Closure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main Group: This an observational registry - there is only one group

SUMMARY:
Canadian WATCHMAN Registry is a multicentre (8 Centres) Canadian prospective, non-randomized, registry to enrol 100 consecutive patients undergoing LAA closure with the WATCHAN device to study the safety and effectiveness of the WATCHMAN device

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia with current prevalence estimated at 1.5-2% of the general population. AF is a major cause of stroke, responsible for 15% of all strokes and 30% of strokes in patients age >80. Stroke is the leading cause of long-term disability and is the 4th leading cause of death in the US. Anticoagulation is the mainstay therapy for preventing strokes in AF with a 64% relative stroke reduction and 26% relative mortality benefit with warfarin therapy. Warfarin or newer anticoagulation treatments (NOAC) have been associated with increased risk of major bleeding and therefore a significant proportion (30-50%) of eligible patients do not receive therapy due to perceived risk of bleeding. The need for newer therapy is therefore required and percutaneous left atrial appendage closure (LAAC) devices have been investigated for patients with high risk of stroke and contra-indication to long term oral anticoagulation therapy. The WATCHMAN device is one of the leading LAA closure devices and with the most world-wide clinical experience. The investigators are running a multicentre (8 Centres) Canadian prospective, non-randomized, registry to enrol 100 consecutive patients undergoing LAA closure with the WATCHAN device to study the safety and effectiveness of the WATCHMAN device.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, and
* CHADS2 ≥1 and/or CHADS-VASc ≥2, and
* Prior major bleeding (intracranial, gastrointestinal bleeding, intraocular, respiratory, genitourinary, retroperitoneal, pericardial, anemia requiring transfusions, etc.), or contraindications to long-term OAC (HASBLED ≥3, high fall risk, cerebral aneurysm, blood dyscrasias, aortic dissection, etc.), or failure of OAC (stroke/TIA while on OAC)

Exclusion Criteria:

* Presence of LAA thrombus
* Severe untreated mitral stenosis (no prior valve replacement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing WATCHMAN device Implantation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events | From up to 24 Months from procedure
  Composite: Cardiovascular death (or unexplained death), device embolization, stroke, systemic embolism, myocardial infarction, cardiac tamponade, major bleeding, and the need for cardiovascular surgery

SECONDARY OUTCOMES:
Long-term Events | From hospital discharge to 24 Months
  Composite: Overall mortality, cardiovascular mortality, ischemic and hemorrhagic stroke, systemic embolization, late device embolization (beyond hospitalization)
Procedural Technical Success | Procedural (up to the end of procedure)
  Procedure duration and complications
Procedural complications | Procedural (up to hospital discharge)
  Stroke (ischemic and hemorrhagic), air embolism, pericardial effusion (minor - not requiring intervention; serious - requiring percutaneous or surgical drainage), cardiac perforation, device embolization, major or life-threatening/disabling bleeding

OTHER OUTCOMES:
Ability to switch to single antiplatelet therapy | up to 3 Months from procedure
Prevalence and severity of residual leak | up to 3 Months from procedure
Prevalence of device thrombus | up to 3 Months from procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Saw, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation: a major contributor to stroke in the elderly. The Framingham Study. Arch Intern Med. 1987 Sep;147(9):1561-4. PMID 3632164
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Zabalgoitia M, Halperin JL, Pearce LA, Blackshear JL, Asinger RW, Hart RG. Transesophageal echocardiographic correlates of clinical risk of thromboembolism in nonvalvular atrial fibrillation. Stroke Prevention in Atrial Fibrillation III Investigators. J Am Coll Cardiol. 1998 Jun;31(7):1622-6. doi: 10.1016/s0735-1097(98)00146-6. PMID 9626843
- [Background] Hughes M, Lip GY; Guideline Development Group, National Clinical Guideline for Management of Atrial Fibrillation in Primary and Secondary Care, National Institute for Health and Clinical Excellence. Stroke and thromboembolism in atrial fibrillation: a systematic review of stroke risk factors, risk stratification schema and cost effectiveness data. Thromb Haemost. 2008 Feb;99(2):295-304. doi: 10.1160/TH07-08-0508. PMID 18278178
- [Background] Fagan SM, Chan KL. Transesophageal echocardiography risk factors for stroke in nonvalvular atrial fibrillation. Echocardiography. 2000 May;17(4):365-72. doi: 10.1111/j.1540-8175.2000.tb01152.x. PMID 10979009